CLINICAL TRIAL: NCT03788434
Title: CONSORTIUM - A Double-Blind Placebo-Controlled Phase 2 Study of VE303 for Prevention of Recurrent Clostridium (Clostridioides) Difficile Infection
Brief Title: Phase 2 Study of VE303 for Prevention of Recurrent Clostridioides Difficile Infection
Acronym: CONSORTIUM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vedanta Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CONSORTIUM (VE303-002)
Record Dates: First submitted 2018-12-19; First posted 2018-12-27 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Clostridium Difficile Infection Recurrence; Clostridium Difficile Infection; Clostridium Difficile; Clostridioides Difficile Infection Recurrence; Clostridioides Difficile Infection; Clostridioides Difficile; CDI
Keywords: Clostridium Difficile Infection Recurrence; Clostridium Difficile Infection; Clostridium Difficile; VE303; Consortium; Vedanta; CDI; C. Diff; CDiff; Clostridiodes Difficile Infection Recurrence; Clostridiodes Difficile Infection; Clostridioides Difficile
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Intervention Model Description: This Phase 2 study evaluated the safety and efficacy of the study drug, VE303, at preventing subsequent CDI-associated diarrhea compared with placebo, following completion of at least 1 successful course of SOC antibiotics for subjects with pCDI at high risk for recurrence or subjects with rCDI.
  Participants in the study were randomized into 3 arms in a 1:1:1 ratio of high dose VE303, low dose VE303, and placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To reduce potential bias and increase study data integrity, study participants, care providers, site investigators, and study outcomes assessors were masked to study treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VE303 High Dose (Experimental): Study subjects assigned the high dose VE303 arm took 10 capsules (dosage: 8.0 × 10^9 CFU daily) containing VE303 per day for 14 days.
  Interventions: Drug: VE303
- VE303 Low Dose (Experimental): Study subjects assigned to the low dose VE303 arm took 2 capsules (dosage: 1.6 × 10^9 CFU daily) containing VE303 per day for 14 days.
  Interventions: Drug: VE303
- Placebo (Placebo Comparator): Study subjects assigned to the placebo dose arm took placebo capsules each day for 14 days. The capsules did not contain any VE303.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VE303 — VE303 is a live biotherapeutic product containing 8 clonal human commensal bacterial strains manufactured under Good Manufacturing Practices (GMP) conditions.
  Arms: VE303 High Dose; VE303 Low Dose
Drug: Placebo — Placebo capsules contained microcrystalline cellulose and were visually identical to VE303 capsules. Placebo capsules did not contain any VE303 Drug Product.
  Arms: Placebo

SUMMARY:
This study evaluated the safety and efficacy of VE303 for participants with primary C. difficile infection (pCDI) at high risk for recurrence or subjects with recurrent C. difficile infections (rCDI).

DETAILED DESCRIPTION:
CONSORTIUM was a randomized, placebo-controlled double-blind Phase 2 study to evaluate safety, tolerability, pharmacokinetics/pharmacodynamics, and efficacy of VE303 in prevention of subsequent Clostridioides difficile infection (CDI) -associated diarrhea compared with placebo following completion of at least 1 successful course of standard-of-care (SOC) antibiotics. VE303 or placebo capsules were taken orally for 14 days after completion of a course of SOC antibiotics. The proportions of subjects experiencing a confirmed CDI recurrence within 8 weeks after the first dose of study treatment were compared across the study arms, to understand the efficacy of VE303 in preventing rCDI.

The study originally planned to enroll 146 subjects but through a protocol amendment was revised to an enrollment target of 60 to 80 subjects with a prior history of CDI diarrhea or first occurrence of CDI diarrhea with a higher risk for recurrence. Subjects must have had a positive C. difficile stool sample and have responded to SOC antibiotic treatment.

ELIGIBILITY:
Partial Inclusion Criteria:

1. Able and willing to provide written informed consent
2. Subjects with a qualifying CDI episode who had a prior history of CDI diarrhea (≥ 18 years of age) or first occurrence of CDI diarrhea with a higher risk for recurrence (≥ 75 years of age, or ≥ 65 years of age with one or more prespecified conditions)
3. CDI symptoms must have started within 30 days (inclusive) prior to the day of randomization
4. The diarrhea was considered unlikely to have another etiology.
5. Completed an Investigator's choice SOC antibiotic regimen of a minimum of 10 days and up to 21 days of total duration
6. Have a positive C. difficile stool
7. Recovered from any complications of severe or fulminant CDI and clinically stable by the time of randomization.

Partial Exclusion Criteria:

1. History of diarrhea (defined as 3 or more loose stools per day lasting for at least 4 weeks) that was not related to C. difficile infection within the 3 months prior to randomization.
2. Known or suspected toxic megacolon and/or known small bowel ileus at the time of randomization.
3. Contraindication to oral/enteral therapy (e.g., severe reflux, severe nausea/vomiting, or ileus).
4. Prior administration of genetically modified investigational live bacterial/fungal/bacteriophage/viral isolates for CDI-associated diarrhea
5. History of administration of fecally-derived investigational live biotherapeutic products, or fecally-derived live bacterial isolates for CDI-associated diarrhea including fecal microbiota transplantation (FMT) within the last 6 months.
6. Use of drugs that alter gut motility
7. History of acute leukemia or hematopoietic stem cell transplantation or myelosuppressive chemotherapy within 2 months prior to randomization.
8. Subjects with compromised immune system
9. Major gastrointestinal surgery (e.g., significant bowel resection or diversion) within 3 months prior to randomization or any history of total colectomy or bariatric surgery that disrupts the gastrointestinal lumen.
10. History of confirmed celiac disease, inflammatory bowel disease, short gut, gastrointestinal tract fistulas, or ischemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darrell Pardi, MD, Principal Investigator — Mayo Clinic
Locations (37):
- United States (29):
  - Phoenix Clinical, LLC, Phoenix, Arizona
  - Mayo Clinic, Clinical Studies Unit, Phoenix, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Alliance Research Institute, Canoga Park, California
  - University of California, Davis Medical Center, Sacramento, California
  - Ventura Clinical Trials, Ventura, California
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Innovative Research of West Florida, Clearwater, Florida
  - Gastro Florida, Clearwater, Florida
  - University of Florida, Gainesville, Florida
  - Guardian Angel Research Center, Tampa, Florida
  - Anne Arundel Health System Research Insitute, Annapolis, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Covenant HealthCare, Saginaw, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - New York University Langone Medical Center, New York, New York
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Toledo Institute of Clinical Research Inc, Toledo, Ohio
  - TruCare Internal Medicine and Infectious Diseases, DuBois, Pennsylvania
  - Frontier Clinical Research, LLC, Uniontown, Pennsylvania
  - Advanced Clinical Research-Be Well MD, Cedar Park, Texas
  - Texas Centers for Infectious Disease Associates, Fort Worth, Texas
  - Clinrx Research Joseph INC, Plano, Texas
  - Infectious Disease Associates of Central Virginia Infectious Disease, Lynchburg, Virginia
  - Seattle Infectious Disease Clinic, Seattle, Washington
  - Advanced Clinical Research-Spokane Gastroenterology, Spokane, Washington
- Canada (8):
  - Foothills Medical Centre - Microbial Health Clinic, Calgary, Alberta
  - CARe Clinic, Red Deer, Alberta
  - Moncton Hospital, Moncton, New Brunswick
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Viable Clinical Research, Scarborough Village, Ontario
  - Q&T Research Chicoutimi, Chicoutimi, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
  - Centre intégré universitaire de santé et de services sociaux de la Mauricie-et-, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Louie T, Golan Y, Khanna S, Bobilev D, Erpelding N, Fratazzi C, Carini M, Menon R, Ruisi M, Norman JM, Faith JJ, Olle B, Li M, Silber JL, Pardi DS. VE303, a Defined Bacterial Consortium, for Prevention of Recurrent Clostridioides difficile Infection: A Randomized Clinical Trial. JAMA. 2023 Apr 25;329(16):1356-1366. doi: 10.1001/jama.2023.4314. PMID 37060545

RESULTS

PARTICIPANT FLOW:
Groups:
- VE303 High Dose: Study subjects assigned to the high dose VE303 arm took 10 capsules containing VE303 per day for 14 days.
  VE303: VE303 is a live biotherapeutic product containing 8 clonal human commensal bacterial strains manufactured under GMP conditions.
- VE303 Low Dose: Study subjects assigned to the low dose VE303 arm took 2 capsules containing VE303 per day for 14 days.
  VE303: VE303 is a live biotherapeutic product containing 8 clonal human commensal bacterial strains manufactured under GMP conditions.
- Placebo: Study subjects assigned to the placebo dose arm took placebo capsules each day for 14 days. The capsules did not contain any VE303.
  Placebo: Placebo capsules contained microcrystalline cellulose and were visually identical to VE303 capsules.
Period: Overall Study
Arm/Group | VE303 High Dose | VE303 Low Dose | Placebo
Started | 30 | 27 | 22
Completed | 29 | 27 | 22
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VE303 High Dose | VE303 Low Dose | Placebo | Total
Number analyzed (Participants) | 30 | 27 | 22 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 12 | 12 | 40
  >=65 years | 14 | 15 | 10 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (14.99) | 62.9 (17.85) | 60.8 (15.98) | 62.1 (16.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 17 | 56
  Male | 11 | 7 | 5 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 28 | 27 | 22 | 77
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 29 | 25 | 22 | 76
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 14 | 49
  Canada | 12 | 10 | 8 | 30

OUTCOME MEASURES:

1. Primary Outcome: CDI Recurrence Week 8
Description: Percentage of participants with toxin-positive, laboratory-confirmed, or clinically diagnosed and treated CDI recurrence before or at Week 8 (i.e., 8 weeks after the first dose of study treatment).
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | VE303 High Dose | VE303 Low Dose | Placebo
Number analyzed (Participants) | 29 | 27 | 22
Participants
  C. difficile recurrences (toxin-positive) | 4 | 9 | 5
  C. difficile recurrences (laboratory-confirmed) | 4 | 10 | 8
  C. difficile recurrences (laboratory-confirmed or clinically diagnosed and treated) | 4 | 10 | 10

2. Secondary Outcome: VE303 Strains Detected
Description: Characterize the number of VE303 strains detected in the fecal microbiome at week 24.
Time Frame: 24 weeks
Population: Enrolled subjects who provided stool samples for analysis at week 24.
Measure: Mean (Standard Deviation); unit: Number of VE303 strains detected
Arm/Group | VE303 High Dose | VE303 Low Dose | Placebo
Number analyzed (Participants) | 20 | 21 | 14
Number of VE303 strains detected | 3.25 (2.807) | 1.62 (1.962) | 0.36 (0.633)

3. Secondary Outcome: VE303 Relative Abundance
Description: Proportion of VE303 strains is defined as the abundance proportion of all 8 VE303 strains relative to the total microbial composition of the sample.
Time Frame: 24 weeks
Population: Enrolled subjects who provided stool samples for analysis at week 24.
Measure: Mean (Standard Deviation); unit: Proportion of VE303 strains
Groups:
- VE303 High Dose: Study subjects assigned the high dose VE303 arm took 10 capsules containing VE303 per day for 14 days.
  VE303: VE303 is a live biotherapeutic product containing 8 clonal human commensal bacterial strains manufactured under GMP conditions.
Arm/Group | VE303 High Dose | VE303 Low Dose | Placebo
Number analyzed (Participants) | 20 | 21 | 14
Proportion of VE303 strains | 0.01186 (0.013897) | 0.00775 (0.016007) | 0.00097 (0.002297)

4. Other Pre Specified Outcome: CDI Recurrence Week 4
Description: Percentage of participants with toxin-positive, laboratory-confirmed, or clinically diagnosed and treated CDI recurrence before or at Week 4 (i.e., 4 weeks after the first dose of study treatment).
Time Frame: 4 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | VE303 High Dose | VE303 Low Dose | Placebo
Number analyzed (Participants) | 29 | 27 | 22
Participants
  C. difficile recurrences (toxin-positive) | 4 | 9 | 2
  C. difficile recurrences (laboratory-confirmed) | 4 | 10 | 5
  C. difficile recurrences (laboratory-confirmed, or clinically diagnosed and treated) | 4 | 10 | 6

5. Other Pre Specified Outcome: CDI Recurrence Week 12
Description: Percentage of participants with toxin-positive, laboratory-confirmed, or clinically diagnosed and treated CDI recurrence before or at Week 12 (i.e., 12 weeks after the first dose of study treatment).
Time Frame: 12 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | VE303 High Dose | VE303 Low Dose | Placebo
Number analyzed (Participants) | 29 | 27 | 22
Participants
  C. difficile recurrences (toxin-positive) | 4 | 9 | 5
  C. difficile recurrences (laboratory-confirmed) | 4 | 10 | 8
  C. difficile recurrences (laboratory-confirmed, or clinically diagnosed and treated) | 4 | 10 | 10

6. Other Pre Specified Outcome: CDI Recurrence Week 24
Description: Percentage of participants with toxin-positive, laboratory-confirmed, or clinically diagnosed and treated CDI recurrence before or at Week 24 (i.e., 24 weeks after the first dose of study treatment).
Time Frame: 24 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | VE303 High Dose | VE303 Low Dose | Placebo
Number analyzed (Participants) | 29 | 27 | 22
Participants
  C. difficile recurrences (toxin-positive) | 4 | 9 | 5
  C. difficile recurrences (laboratory-confirmed) | 5 | 11 | 8
  C. difficile recurrences (laboratory-confirmed or clinically diagnosed and treated) | 5 | 11 | 10

7. Other Pre Specified Outcome: Microbiota Diversity
Description: Characterize the fecal microbiome Shannon Diversity at week 24.
Time Frame: 24 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Determine the Recommended VE303 Phase 3 Dose Regimen(s).
Description: Determine the recommended VE303 phase 3 dose regimen(s) based on safety and efficacy, as indicated by the CDI recurrence rate for the duration of the study.
Time Frame: 31 Months 1 Week
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Changes in the Fecal Metabolomic Profile, Including Short-chain Fatty Acids and Bile Acids.
Description: Changes in the fecal metabolomic profile, including short-chain fatty acids and bile acids for the duration of the study.
Time Frame: 31 Months 1 Week
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Taxonomic Composition
Description: Characterize Taxonomic Composition
Time Frame: 31 Months, 1 Week
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | VE303 High Dose | VE303 Low Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/27 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/29 | 4/27 | 2/22
Other Adverse Events (participants affected / at risk) | 28/29 | 27/27 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VE303 High Dose (N=29) | VE303 Low Dose (N=27) | Placebo (N=22)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CDI (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Transfusion Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VE303 High Dose (N=29) | VE303 Low Dose (N=27) | Placebo (N=22)
Diarrhea (Gastrointestinal disorders) | 21 (243) | 23 (213) | 19 (114)
Nausea (Gastrointestinal disorders) | 6 (7) | 6 (6) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 5 (7) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (2) | 4 (4) | 3 (3)
Abdominal Distension (Gastrointestinal disorders) | 2 (3) | 1 (2) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 2 (2) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 4 (4) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 2 (2)
Malaise (General disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Blood Potassium Increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (3) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT03788434/Prot_002.pdf
  • Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT03788434/SAP_003.pdf